CLINICAL TRIAL: NCT03842124
Title: Improving Safety of Lead Extraction Procedures by Traction Force Sensing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Siva Mulpuru, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-007322
Record Dates: First submitted 2019-01-09; First posted 2019-02-15 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Implantable Electronic Device Infection; Cardiovascular Infections
Keywords: infection; pacemaker; ICD; CRT
MeSH Terms: conditions — Cardiovascular Infections; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is randomized such that the same operator can be doing the extraction with force gauge with or without the force information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Use of bidirectional rail (superior and inferior approaches) and force sensing using a force gauge to optimize Force application to less than 8 lbs during the extraction procedure.
  Interventions: Other: Force gauge
- Control (No Intervention): Conventional lead extraction procedures using a superior approach is performed by experienced operators. Although force information is available the operators are blinded to the information. Inferior rail is left to the discretion of the operator.

INTERVENTIONS:
Other: Force gauge — The investigators postulate that use of bidirectional traction (superior and inferior directions) and feedback from a digital force gauge is associated with minimal lead displacement compared to conventional lead extraction.
  Arms: Intervention

SUMMARY:
Death and vascular tears occur in up to 1% of the patients undergoing lead extraction procedures. These complications are due to abnormal force vectors during the procedure. The investigators postulate that use of bidirectional traction (superior and inferior directions) and feedback from a digital force gauge is associated with minimal lead displacement compared to conventional lead extraction. Lead displacement is an indirect risk factor for potentially fatal lead extraction complications

DETAILED DESCRIPTION:
Use of force no greater than 8 pounds of tension will improve lead extraction and minimize lead displacement compared to current standard of care methods which do not limit the force applied. Among subjects undergoing lead extraction procedures for CIED infection, bidirectional rail (superior and inferior) and traction force objective feedback using Force gauge is associated with minimal displacement (<1cm) of the leads (surrogate marker) on fluoroscopy compared to conventional lead extraction. • The research nature of the protocol is explicitly explained to the patient and an informed consent is explained obtained from the patient prior to the procedure. Only patients with CIED infections requiring lead extraction are enrolled in the study. Patients are risk stratified based on our current risk stratifications scheme. Multiple superior and inferior venous accesses are obtained during the procedure. The leads are prepared using locking stylets. Baseline fluoroscopic image of the position of the leads is stored. A deflectable sheath and traction forceps are deployed from the groin to provide downward rail in the force feedback arm. Locking stylet from the lead is in turn attached to a Force gauge (McMaster-Carr Santa Fe Springs, CA). The procedure is performed using continuous fluoroscopic image save tool during the procedure for post procedural viewing and analysis. The patients are randomized to the active arm (to keep force around 8 lb) or the control arm (tactile force discretion based on the operator. The investigator is blinded to the force gauge reading for half of the patients enrolled in the study. For the other half of the patients, the operator optimizes the force to prevent overexertion (<8-9 pounds). Three point along the lead course evaluated during the study. Position of downward turn of the lead in the SVC, heel of the lead (only in case of RV lead) and the lead tip positions are evaluated. The investigators postulate that there will be at least 5 cine-fluoroscopic views per every lead. The investigators hypothesize that use of bidirectional rail and force feedback is associated with minimal displacement of the lead on fluoroscopy.

ELIGIBILITY:
Inclusion criteria:

• Patients with CIED infection requiring extraction

Exclusion criteria:

* Age <18 years
* Noninfectious reasons for extraction
* Patients with cognitive impairment, who are unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Fluoroscopic lead displacement | Intra-procedure measurements
  The primary objective of the study is to evaluate the effect of traction force as measured by a digital force gauge on fluoroscopic lead displacement during lead extraction procedures. The investigators hypothesize that the lead displacement on fluoroscopy will be less than 1 cm when the traction force is limited to less than 8 lb.

CONTACTS AND LOCATIONS:
Overall Officials: Siva K Mulpuru, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials